CLINICAL TRIAL: NCT00916500
Title: A Phase II Trial of Concurrent Chemoradiation With Cisplatin Every 3 Week in Advanced Cervical Cancer Patients
Brief Title: Concurrent Chemoradiation With Cisplatin Every 3 Week in Advanced Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Cancer Center Hospital (Other)
Responsible Party: Principal Investigator, Sang-Young Ryu, Chair of Cerivcal/Ovarian Cancer Center, Korea Cancer Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCCH GY 1001
Record Dates: First submitted 2009-06-07; First posted 2009-06-09 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: CERVICAL NEOPLASMS
Keywords: CERVICAL CANCER, CONCURRENT CHEMORADIATION, CISPLATIN
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CISPLATIN (Experimental): Patients With Locally Advanced Cervical Cancer Who Underwent Concurrent Chemoradiation; Cisplatin 75mg/m2 IV Every 3 Week For 3 Cycles; External Pelvic Radiation 40 Gy; Brachytherapy Up to 85-90 Gy To Point A
  Interventions: Drug: CONCURRENT CHEMORADIATION (CISPLATIN)

INTERVENTIONS:
Drug: CONCURRENT CHEMORADIATION (CISPLATIN) — Cisplatin IV 75mg/m2 Every 3 Week For 3 Cycles; External Pelvic Radiation 40Gy; Brachytherapy Up To 85-90 Gy To Point A
  Other Names: Cisplatin

SUMMARY:
Concurrent chemoradiation (CCRT) is the standard therapy for locally advanced cervical cancer.

However, the most effective chemotherapy regimen is controversial. Weekly cisplatin, hydroxyurea + cisplatin, 5-FU + cisplatin are tested in clinical trials.

Weekly cisplatin needs frequent hospital visits and had a poor compliance profile in korea.

Combination chemotherapy regimens had more adverse effects than weekly cisplatin without improving outcomes.

We conducted a retrospective analysis comparing weekly cisplatin with cisplatin every 3 weeks and observed favorable outcome for cisplatin every 3 weeks regimen (still not published).

Therefore, we designed a phase 2 trial evaluating the efficacy and feasibility of CCRT with cisplatin every 3 weeks.

DETAILED DESCRIPTION:
Cervical carcinoma is one of the most common gynecologic cancers worldwide. The prognosis of cervical cancer is favorable, with an approximately 80-90% 5-year survival rate in early-stage disease. However, advanced disease carries a poor prognosis.

Current standard treatment for locally advanced cervical cancer, which is not eligible for surgical treatment, is cisplatin-based concurrent chemoradiation. On the basis of the results of five randomized clinical trials, which consistently showed improved survival in patients treated with cisplatin-based chemoradiation, the U.S. National Cancer Institute (NCI) announced in 1992 that "Strong consideration should be given to the incorporation of concurrent cisplatin-based chemotherapy with radiotherapy in women who require radiotherapy for treatment of cervical cancer".

Although recently reported meta-analyses also demonstrated improved local control rates and survival with cisplatin-based chemotherapy concurrent with radiation, the optimal cisplatin dose and dosing schedule are still undetermined.

Among the previous five randomized clinical trials, two trials performed by the Gynecologic Oncology Group (GOG) used weekly cisplatin 40 mg/m2 while the other three trials used tri-weekly cisplatin at a dosage range of 50 mg/m2 to 75 mg/m2 combined with 5-fluorouracil (5-FU). Despite the diversity in cisplatin dose and dosing schedules, weekly cisplatin at a dose of 40 mg/m2 concurrent to RT is widely accepted as the standard regimen of CRT because of its convenience, equal effectiveness, and favorable toxicity in comparison to other 5-FU combined regimens.

However weekly cisplatin regimen needs frequent hospital visits and had a poor compliance profile in korea. With weekly cisplatin regimen, planned treatment was not completed in 58% patients adn treatment delayed in 29% patient. among these patients, 9% patients were not related associated toxicities.

To overcome toxicities and poor compliance of weekly regimen, the investigators tried to evaluate the efficacy and feasibility of CCRT with cisplatin 75mg/m2 every 3 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Histologically confirmed cervical cancer
2. Clinical stage from 2b to 4a
3. Equal to or younger than 75
4. Gog performance status 0 - 2
5. Anc > 1500/mm3 and platelet > 100000/mm3 and hemoglobin > 10 g/dl
6. Serum creatinine < 2.0
7. AST, ALT < 3 * upper normal level and serum bilirubin < 1.5 mg/dl
8. Expected survival equal to or longer than 6 months
9. Who agreed to participate in this study

Exclusion criteria:

1. History of chemotherapy or radiation to abdomen or pelvis
2. History of other cancers
3. Pleural or pericardial effusion, ascites causing respiratory difficulties equal to or worse than NCI CTCAE grade 2
4. History of allergy or hypersensitivity reaction to platinum
5. History of atrial or ventricular arrhythmia, or congestive heart failure
6. Uncontrolled diabetes, hypertension, or ischemic heart disease
7. Myocardial infarction within 6 months
8. Sepsis or severe infection
9. Pregnant women
10. An unapproved therapy within 30 days before enrollment
11. Other serious diseases which can threat the safety of participants or impair the ability of participants to participate this trial

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
DISEASE-FREE SURVIVAL | 5 YEAR AFTER THERAPY

SECONDARY OUTCOMES:
DISEASE-FREE SURVIVAL | 2 YEAR AFTER THERAPY
OVERALL SURVIVAL | FROM THERAPY TO DEATH
RECURRENCE RATE | 2 YEAR AFTER THERAPY
RECURRENCE RATE | 5 YEAR AFTER THERAPY

CONTACTS AND LOCATIONS:
Overall Officials: SANG YOUNG RYU, M.D., Principal Investigator — STAFF
Locations (1):
- Korea Cancer Center Hospital, Korea Institute of Radiological & Medical Sciences, Seoul, South Korea